CLINICAL TRIAL: NCT05337527
Title: Neuromuscular Responses to Acute Beetroot Ingestion in Women Older Adults. Performance and Side Effects
Brief Title: Neuromuscular Responses to Acute Beetroot Ingestion in Women Older Adults
Acronym: BEET_ELDERLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Álvaro López Samanés, PhD, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: uFrancisco_Vitoria_
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Dietary Supplement; Placebo
Keywords: dietary supplements; nitrate; neuromuscular function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot supplementation (Experimental): One serving 70 mL of beetroot juice (6.4 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) 3 h before initiating the testing session.
  Interventions: Dietary Supplement: beetroot juice
- Placebo supplementation (Placebo Comparator): One serving 70 mL of beetroot juice placebo (0.04 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) 3 h before initiating the testing session.
  Interventions: Dietary Supplement: beetroot juice

INTERVENTIONS:
Dietary Supplement: beetroot juice — Acute effects of beetroot juice or placebo juice ingestion

SUMMARY:
Beetroot juice supplementation has shown the capacity for provoking different physiological effects (e.g. vasodilation and muscle contraction increments). However, the effects of beetroot juice ingestion on neuromuscular performance in women older adults are barely studied. In this randomized placebo-controlled study, we investigated the effects of beetroot acute supplementation in improving neuromuscular performance in women older adults

DETAILED DESCRIPTION:
Beetroot juice supplementation has shown the capacity for provoking different physiological effects that could affect human performance (e.g. vasodilation and muscle contraction increments). Although this dietary supplement has been commonly used for improving sports performance in recreational or professional athletes, the scientific literature in older adults is scarce. Thus, in our knowledge, no previous studies have analyzed the side effects associated to ingestion in this population group. In this randomized placebo-controlled study, we investigated the effects of beetroot acute supplementation in improving neuromuscular performance and side effects associated with ingestion in women older adults.

ELIGIBILITY:
Inclusion Criteria:

* Women >65 or <85 years of age.
* In good health, as determined by the investigator's review of history.

Exclusion Criteria: (based in previous studies on this topic (doi: 10.1093/gerona/glaa311).

Men and women <65 or >85 years of age Unable to provide informed consent Current smokers Significant orthopedic limitations or other contraindications to strenuous exercise Those taking proton pump inhibitors, antacids, xanthine oxidase inhibitors, or on hormone replacement therapy Those taking anti-coagulants or on anti-platelet therapy History of neuromuscular disease (e.g., cervical spondylotic radiculomyelpathy, lumbar spondylosis, amyotrophic lateral sclerosis, Guillain-Barré syndrome, and acquired demyelinating polyneuropathies) Cardiovascular disease (e.g., > stage I hypertension, heart failure, myocardial infarction/ischemia significant myocardial or pericardial diseases (e.g. amyloidosis, constriction), Moderate or severe valvular disease, renal disease, liver disease, or anemia

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Only women older adults were selected for this study.
Enrollment: 9 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Changes in maximal isometric handgrip strength (N) | 1-week
  Using a dynamometer and measuring dominant/ non-dominant side
Changes in 6-m gait speed test | 1-week
  Using a photocell timing gates (seconds)
Changes in Time Up and Go test | 1-week
  Using a photocell timing gates (seconds)
Changes in Sit and Stand Test | 1-week
  Using Power Frail APP
6-Minute Walk Test | 1-week

SECONDARY OUTCOMES:
Rate of perception effort (RPE) | 1-week
  Using a validated scale (1-10 points)
Side effects questionnarie | 1-week
  Using a side-effects questionnarie (YES/NO scale)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro López Samanes, PhD, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No